CLINICAL TRIAL: NCT03467048
Title: Comparison of McGrath Videolaryngoscopy and Direct Laryngoscopy for Intubation in Patients With Morbid Obesity in Non-cardiac Surgery
Brief Title: McGrath Videolaryngoscopy and Direct Laryngoscopy in Morbidly Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-077
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- McGrath videolaryngoscopy (Experimental): Endotracheal intubation using McGrath videolaryngoscopy in an appropriate size (usually blade size 3 or 4)
  Interventions: Device: McGrath videolaryngoscopy
- Direct laryngoscopy (Active Comparator): Endotracheal intubation using direct laryngoscopy with an appropriately sized Macintosh blade (usually size 3 or 4)
  Interventions: Device: Direct laryngoscopy

INTERVENTIONS:
Device: McGrath videolaryngoscopy — Intubations will be performed with a regular endotracheal tube of adequate diameter, usually 7.5 mm or 8.0 mm. Endotracheal tubes will be equipped with a hockey-stick-shaped stylette, which will be prepared by the anesthesiologist in advance.
  The McGrath or the Macintosh blade will be introduced into oral cavity according to manufacturer recommendations and clinical practice. Minor airway manipulation procedures including BURP or Sellick maneuvers will be allowed to improve visualization of the vocal cords.
  Arms: McGrath videolaryngoscopy
Device: Direct laryngoscopy — Intubations will be performed with a regular endotracheal tube of adequate diameter, usually 7.5 mm or 8.0 mm. Endotracheal tubes will be equipped with a hockey-stick-shaped stylette, which will be prepared by the anesthesiologist in advance.
  The McGrath or the Macintosh blade will be introduced into oral cavity according to manufacturer recommendations and clinical practice. Minor airway manipulation procedures including BURP or Sellick maneuvers will be allowed to improve visualization of the vocal cords.
  Arms: Direct laryngoscopy

SUMMARY:
Our goal is to compare conventional direct laryngoscopy using a Macintosh blade with the McGrath videolaryngoscope for endotracheal intubation in very morbidly obese patients undergoing non-cardiac surgery. Specifically, we propose to test the primary hypotheses that videolaryngoscopy improves visualization of the vocal cords, defined with modified Cormack and Lehane classification, compared to direct laryngoscopy.

DETAILED DESCRIPTION:
In the preoperative period, patient's airway data will be recorded by a research coordinator or anesthesia provider (Table 1). Patients will be positioned supine and in a standardized ramped position on the OR table. Patients will be pre-medicated with midazolam 0-2 mg IV, as clinically appropriate. All patients will be pre-oxygenated until the fraction of expired oxygen exceeds 80%. General anesthesia will be induced as preferred by the attending anesthesiologist, usually with a combination of lidocaine 1 mg/kg, propofol 2-5 mg/kg, fentanyl 1-3 µg/kg, and rocuronium 0.6-1.2 mg/kg or succinylcholine 1.5 mg/kg.

Manual bag-mask ventilation will be initiated, with no restriction on the use of oral airways, nasal airways, laryngeal masks. Complete muscle relaxation will be confirmed by absence of palpable twitches in response to supra-maximal train-of-four stimulation of the ulnar nerve at the wrist. After confirming adequate bag mask manual ventilation, patients will be randomized 1:1, stratified for BMI >50 kg/m2, to:

* Direct laryngoscopy using an appropriately sized Macintosh blade (usually size 3 or 4);
* McGrath videolaryngoscopy in an appropriate size (usually blade size 3 or 4). Randomization will be based on computer-generated codes accessed from the Redcap system shortly before anesthetic induction. Allocation will thus be concealed until the last possible minute.

Intubations will be performed with a regular endotracheal tube of adequate diameter, usually 7.5 mm or 8.0 mm. Endotracheal tubes will be equipped with a hockey-stick-shaped stylette, which will be prepared by the anesthesiologist in advance.

The McGrath or the Macintosh blade will be introduced into oral cavity according to manufacturer recommendations and clinical practice. Minor airway manipulation procedures including BURP or Sellick maneuvers will be allowed to improve visualization of the vocal cords.

If initial intubation attempts fails, the endotracheal tube will be removed and manual bag mask ventilation will resume. Minor adjustments of patient's position and/or tube stylette are allowed as clinically appropriate. Up to three intubation attempts will be made as necessary. Further airway management will follow clinical assessment of the anesthesiologist. Additionally, throughout the procedure, the anesthesiologist could terminate the study participation.

Once intubation is achieved, the endotracheal tube will be connected to the anesthesia circuit. Mechanical ventilation with O2 and air will be adjusted to maintain end-tidal PCO2 between 32 and 35 mmHg as clinically necessary. Maintenance of general anesthesia will be provided, as clinically indicated.

At the end of the surgical procedure, patients will be extubated and transferred to the post anesthesia care unit (PACU). Patients will then be assessed for postoperative complications 2 hours following extubation, either in the PACU or surgical ward.

Measurements Table 1. Demographic and morphometric characteristics will be collected from electronic medical records.

1. Age
2. Gender
3. Race
4. BMI
5. ASA status
6. Charlson score
7. Smoking status
8. Airway examination

   1. History of obstructive sleep apnea (yes/no)
   2. History of snoring (yes/no)
   3. History of CPAP (yes/no)
   4. History of difficult airway (yes/no)
   5. Mobility of cervical spine (cm)
   6. Mouth opening (cm)
   7. Inter-incisor gap (cm)
   8. Mandibular protrusion test
   9. Thyro-mental distance (cm)
   10. Sterno-mental distance (cm)
   11. Neck circumference (cm)
   12. Upper lip bite test (Class I, II, III)
   13. Mallampati score (1/2/3/4)
   14. Teeth status, Gap/missing teeth, Denture (n)

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery requiring oral endotracheal intubation for general anesthesia;
* Anticipated extubation in the operating room;
* American Society of Anesthesiologists (ASA) physical status 1-3;
* Age between 18 and 99 years;
* Body Mass index ≥ 40 kg/m2.

Exclusion Criteria:

* Refusal of participation by attending anesthesiologist;
* Indicated rapid sequence induction for any reason including, but not limited to high risk of aspiration
* Indicated fiberoptic awake intubation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ruetzler K, Rivas E, Cohen B, Mosteller L, Martin A, Keebler A, Maheshwari K, Steckner K, Wang M, Praveen C, Khanna S, Makarova N, Sessler DI, Turan A. McGrath Video Laryngoscope Versus Macintosh Direct Laryngoscopy for Intubation of Morbidly Obese Patients: A Randomized Trial. Anesth Analg. 2020 Aug;131(2):586-593. doi: 10.1213/ANE.0000000000004747. PMID 32175948

RESULTS

PARTICIPANT FLOW:
Groups:
- McGrath Videolaryngoscopy: Endotracheal intubation using McGrath videolaryngoscopy in an appropriate size (usually blade size 3 or 4)
  McGrath videolaryngoscopy: Intubations will be performed with a regular endotracheal tube of adequate diameter, usually 7.5 mm or 8.0 mm. Endotracheal tubes will be equipped with a hockey-stick-shaped stylette, which will be prepared by the anesthesiologist in advance.
  The McGrath or the Macintosh blade will be introduced into oral cavity according to manufacturer recommendations and clinical practice. Minor airway manipulation procedures including BURP or Sellick maneuvers will be allowed to improve visualization of the vocal cords.
- Direct Laryngoscopy: Endotracheal intubation using direct laryngoscopy with an appropriately sized Macintosh blade (usually size 3 or 4)
  Direct laryngoscopy: Intubations will be performed with a regular endotracheal tube of adequate diameter, usually 7.5 mm or 8.0 mm. Endotracheal tubes will be equipped with a hockey-stick-shaped stylette, which will be prepared by the anesthesiologist in advance.
  The McGrath or the Macintosh blade will be introduced into oral cavity according to manufacturer recommendations and clinical practice. Minor airway manipulation procedures including BURP or Sellick maneuvers will be allowed to improve visualization of the vocal cords.
Period: Overall Study
Arm/Group | McGrath Videolaryngoscopy | Direct Laryngoscopy
Started | 66 | 64
Completed | 66 | 63
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | McGrath Videolaryngoscopy | Direct Laryngoscopy | Total
Number analyzed (Participants) | 66 | 63 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (14) | 47 (13) | 49 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 46 | 95
  Male | 17 | 17 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 54 | 53 | 107
  Race: African American | 9 | 9 | 18
  Race: Hispanic | 2 | 1 | 3
  Race: Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 66 | 63 | 129

OUTCOME MEASURES:

1. Primary Outcome: Classification of Glottis Visualization
Description: Glottis visualization is evaluated according to the modified Cormack and Lehane classification. It is a grading system from 1 to 4: 1 = full view of glottis; 2a = partial view of glottis;2b = only posterior extremity of glottis seen or only arytenoid cartilages; 3 = only epiglottis seen, none of glottis seen; 4 = neither glottis nor epiglottis seen.
Time Frame: At intubation
Measure: Count of Participants; unit: Participants
Arm/Group | McGrath Videolaryngoscopy | Direct Laryngoscopy
Number analyzed (Participants) | 66 | 63
Participants
  1 | 45 | 23
  2a | 11 | 16
  2b | 7 | 14
  3 | 3 | 6
  4 | 0 | 4
Statistical Analysis 1: Comparison: McGrath Videolaryngoscopy vs Direct Laryngoscopy; Test type: Non-Inferiority — Null hypothesis: McGrath Video Laryngoscopy is non-inferior to Macintosh direct laryngoscopy; p < 0.01, t-test, 1 sided; Odds Ratio (OR) = 4.65, 95% CI 2-sided [2.22 to 9.75]

2. Secondary Outcome: Number of Intubation Failure
Description: intubation failure
Time Frame: intubation
Measure: Count of Participants; unit: Participants
Arm/Group | McGrath Videolaryngoscopy | Direct Laryngoscopy
Number analyzed (Participants) | 66 | 63
Participants | 2 | 5
Statistical Analysis 1: Comparison: McGrath Videolaryngoscopy vs Direct Laryngoscopy; Test type: Non-Inferiority — Null hypothesis: McGrath videolaryngoscopy is non-inferior to Direct laryngoscopy; p = 0.08, t-test, 1 sided; Odds Ratio (OR) = 0.3, 0.975% CI 2-sided [0.04 to 2.28]

3. Secondary Outcome: Number of Intubation Attempts Among Those With Successful Intubation
Time Frame: intubation
Population: excluded intubation failure
Measure: Count of Participants; unit: Participants
Arm/Group | McGrath Videolaryngoscopy | Direct Laryngoscopy
Number analyzed (Participants) | 64 | 58
Participants
  1 intubation attempt | 61 | 56
  2 intubation attempts | 3 | 2
Statistical Analysis 1: Comparison: McGrath Videolaryngoscopy vs Direct Laryngoscopy; Test type: Non-Inferiority — Null hypothesis: McGrath videolaryngoscopy is non-inferior to Direct laryngoscopy; p = 0.41, t-test, 1 sided; Odds Ratio (OR) = 0.87, 97.5% CI 2-sided [0.1 to 7.77]

ADVERSE EVENTS:
Time Frame: 6months
Arm/Group | McGrath Videolaryngoscopy | Direct Laryngoscopy
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/63
Other Adverse Events (participants affected / at risk) | 0/66 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT03467048/Prot_SAP_001.pdf